CLINICAL TRIAL: NCT03354663
Title: Multi-Center Acute Safety Trial of TactiCath™ Contact Force Ablation Catheter, Sensor Enabled™ (TactiCath SE) for the Treatment of Drug Refractory Recurrent Symptomatic Paroxysmal Atrial Fibrillation
Brief Title: TactiSense IDE Trial of TactiCath SE for Paroxysmal Atrial Fibrillation
Acronym: TactiSense
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJM-CIP-10216
Record Dates: First submitted 2017-11-17; First posted 2017-11-28 (Actual); Results first posted 2019-08-20 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: paroxysmal atrial fibrillation; PAF; ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- TactiCath SE (Experimental): Catheter ablation with the TactiCath SE ablation catheter to achieve pulmonary vein isolation.
  Interventions: Device: TactiCath SE

INTERVENTIONS:
Device: TactiCath SE — Ablation to achieve pulmonary vein isolation.

SUMMARY:
This clinical investigation is intended to demonstrate the acute safety and effectiveness of ablation with the TactiCath™ Contact Force Ablation Catheter, Sensor Enabled™ (TactiCath SE) for the treatment of drug refractory recurrent symptomatic paroxysmal atrial fibrillation (PAF). This clinical investigation will be conducted under an investigational device exemption (IDE) and is intended to support market approval of the TactiCath SE ablation catheter in the United States. One hundred fifty six (156) subjects will be enrolled at up to 35 investigational sites in the US, Europe, and Australia. This clinical investigation is sponsored by Abbott.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm clinical trial to demonstrate the acute safety and effectiveness of the TactiCath SE catheter for the treatment of PAF against a performance goal. One hundred fifty six (156) subjects will be enrolled at up to 35 investigational sites in the US, Europe, and Australia. Only sites that enroll at least one subject will be part of the analysis population. No center may contribute more than 20% of the total number of enrollments without sponsor pre-approval to exceed this proportion and at least 50% of subjects must be from the United States.

ELIGIBILITY:
Inclusion Criteria:

* Plans to undergo a catheter ablation procedure due to symptomatic PAF that is refractory or intolerant to at least one Class I or III antiarrhythmic drug
* Physician's note indicating recurrent self-terminating AF
* One electrocardiographically documented AF episode within 6 months prior to the index ablation procedure
* At least 18 years of age
* Able and willing to comply with all trial requirements
* Informed of the nature of the trial, agreed to its provisions and has provided written informed consent as approved by the Institutional Review Board/Ethics Committee (IRB/EC) of the respective clinical trial site.

Exclusion Criteria:

* Persistent or long-standing persistent atrial fibrillation (AF)
* Four or more cardioversions in the past 12 months
* Active systemic infection
* Known presence of cardiac thrombus
* Implanted with implantable cardiac defibrillator (ICD)
* Arrhythmia due to reversible causes including thyroid disorders, acute alcohol intoxication, and other major surgical procedures in the preceding 3 months
* Myocardial infarction (MI), acute coronary syndrome, percutaneous coronary intervention (PCI), or valve or coronary bypass grafting surgery within preceding 3 months
* Left atrial diameter > 5.0 cm
* Left ventricular ejection fraction < 35%
* New York Heart Association (NYHA) class III or IV
* Previous left atrial surgical or catheter ablation procedure
* Left atrial surgical procedure or incision with resulting scar
* Previous tricuspid or mitral valve replacement or repair
* Heart disease in which corrective surgery is anticipated within 6 months
* Bleeding diathesis or suspected procoagulant state
* Contraindication to long term antithromboembolic therapy
* Presence of any condition that precludes appropriate vascular access
* Renal failure requiring dialysis
* Known sensitivity to contrast media (if needed during the procedure) that cannot be controlled with pre-medication
* Severe pulmonary disease (e.g., restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces severe chronic symptoms
* Pregnant or nursing
* Presence of other anatomic or comorbid conditions that, in the investigator's opinion, could limit the patient's ability to participate in the clinical trial or to comply with follow up requirements, or impact the scientific soundness of the clinical trial results
* Patient is currently participating in another clinical trial or has participated in a clinical trial within 30 days prior to screening that may interfere with this clinical trial
* Patient is unlikely to survive the protocol follow up period of 12 months
* Body mass index > 40 kg/m2
* Vulnerable subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2019-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Ruffner, PhD MBA, Study Director — Abbott
Locations (21):
- United States (14):
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Scripps Health, La Jolla, California
  - Sequoia Hospital, Redwood City, California
  - South Denver Cardiology Associates, P.C., Littleton, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Florida Hospital, Orlando, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Central Baptist Hospital, Lexington, Kentucky
  - Mayo Clinic, Rochester, Minnesota
  - New York University Hospital, New York, New York
  - Mount Sinai Hospital, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Cardiac Arrhythmia, Austin, Texas
- Australia (3):
  - Ashford Hospital, Adelaide
  - Royal Adelaide Hospital, Adelaide
  - Royal Melbourne Hospital - City Campus, Melbourne
- Germany (2):
  - Herzzentrum Leipzig GmbH, Leipzig, Saxony
  - Herzzentrum Dresden GmbH Universitätsklinik, Dresden
- Italy (2):
  - Ospedale San Raffaele, Milan, Lombardy
  - Centro Cardiologico Monzino, Milan

RESULTS

PARTICIPANT FLOW:
Period: Enrollment to Catheter Insertion
Arm/Group | TactiCath SE
Started | 156
Completed | 151
Not Completed | 5
Not completed — Did not meet inc/exc criteria | 4
Not completed — Adverse Event | 1
Period: Completed 30-day Visit
Arm/Group | TactiCath SE
Started | 151
Completed | 149
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Missed Visit | 1

BASELINE CHARACTERISTICS:
Population: Population includes all subjects with device inserted into vasculature.
Arm/Group | TactiCath SE
Number analyzed (Participants) | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 75
  >=65 years | 76
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65.0 [56.0 to 71.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 125
  Unknown or Not Reported | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 123
  More than one race | 3
  Unknown or Not Reported | 21
Region of Enrollment [Number; unit: participants]
  United States | 101
  Italy | 12
  Australia | 22
  Germany | 21
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.0 (5.0)
Coronary Artery Disease [Count of Participants; unit: Participants] | 20
Heart Failure [Count of Participants; unit: Participants] | 4
Hypertension [Count of Participants; unit: Participants] | 80
Diabetes [Count of Participants; unit: Participants] | 15
Stoke/Transient Ischemic Attack [Count of Participants; unit: Participants] | 14
Myocardial Infarction [Count of Participants; unit: Participants] | 6
Obstructive Sleep Apnea [Count of Participants; unit: Participants] | 20
Structural Heart Disease [Count of Participants; unit: Participants] | 5
Known Family History of Cardiovascular Disease [Count of Participants; unit: Participants] | 81
Left Ventricular Ejection Fraction [Median (Inter-Quartile Range); unit: %] | 60.7 [55.0 to 65.0]
Left Atrium Diameter [Median (Inter-Quartile Range); unit: centimeters] | 3.8 [3.3 to 4.3]
Pacemaker or Implantable Cardiac Monitor [Count of Participants; unit: Participants] | 19

OUTCOME MEASURES:

1. Primary Outcome: Rate of Serious Adverse Events
Description: The primary safety endpoint is the rate of device or procedure-related serious adverse events occurring within 7 days of the index procedure. SAEs related solely to arrhythmia recurrence (without coexisting conditions such as thromboembolism, worsening heart failure, etc.) will not be considered primary safety endpoint events. The SAEs that will be included in this endpoint are:
  * Atrial-esophageal fistula
  * AV block
  * Cardiac Perforation/ Tamponade
  * Death
  * Diaphragmatic paralysis
  * Gastroparesis
  * Hospitalization
  * Myocardial Infarction
  * Pericarditis
  * Pneumothorax
  * Pulmonary edema
  * Pulmonary vein stenosis
  * Stroke
  * Thromboembolism
  * Transient ischemic attack
  * Vascular access complications
  Atrial-esophageal fistula, cardiac perforation/tamponade, and pulmonary vein stenosis that occur >7 days post procedure through 30 days will also contribute to the primary endpoint.
Time Frame: 30 days
Population: All subjects with device inserted into vasculature and either experienced a primary endpoint event or completed 30 days of follow up.
Measure: Count of Participants; unit: Participants
Groups:
- TactiCath SE - Safety Population: Catheter ablation with the TactiCath SE ablation catheter to achieve pulmonary vein isolation.
  TactiCath SE: Ablation to achieve pulmonary vein isolation.
  Includes all subjects with catheter inserted into vasculature.
Arm/Group | TactiCath SE - Safety Population
Number analyzed (Participants) | 149
Participants | 7
Statistical Analysis 1: Comparison: TactiCath SE - Safety Population; The hypothesis is formally expressed as: H0: P ≥ 16.2% Ha: P < 16.2%, where P is the percentage of subjects with a primary safety endpoint event. The hypothesis will be tested based on a one-sided exact test of binomial proportions at the one-sided 0.05 alpha level; Test type: Other — Single arm trial; p < 0.0001, Binomial Exact Test; Proportion = 0.047, 95% CI 1-sided [upper limit 0.0864]

2. Primary Outcome: Number of Participants With Procedural Success
Description: The primary effectiveness endpoint is acute procedural success, where acute procedural success is defined as confirmation of entrance block in all pulmonary veins
Time Frame: 0 days
Population: Effectiveness Population - all subjects with device inserted into vasculature
Measure: Count of Participants; unit: Participants
Arm/Group | TactiCath SE
Number analyzed (Participants) | 151
Participants | 148
Statistical Analysis 1: Comparison: TactiCath SE; Test type: Other — The hypothesis is formally expressed as: H0: P < 90% Ha: P ≥ 90%, where P is the percentage of subjects with acute success. The hypothesis will be tested based on a one-sided exact test of binomial proportions at the one-sided 0.05 alpha level. Rejection of the null hypothesis will indicate study success; p = 0.0001, Binomial Exact Test; Proportion = 0.98, 95% CI 1-sided [lower limit 0.9495]

3. Other Pre Specified Outcome: Average Power Delivered
Description: This outcome is the average power delivered for a case.
Time Frame: During Procedure
Population: The population includes only subjects with at least some radiofrequency energy delivered.
Measure: Median (Inter-Quartile Range); unit: Watts
Groups:
- RF Population: Group of subjects with at least some RF energy delivered
Arm/Group | RF Population
Number analyzed (Participants) | 150
Watts | 29.0 [26.0 to 32.0]

4. Other Pre Specified Outcome: Index Cases Achieving ≥ 90% Lesions With ≥ 10 Contact Force
Description: Proportion of index cases achieving ≥ 90% lesions with ≥10g contact force
Time Frame: 0 days
Population: Population includes all subjects with at least some radiofrequency energy delivered.
Measure: Count of Participants; unit: Participants
Arm/Group | RF Population
Number analyzed (Participants) | 149
Participants | 5

5. Other Pre Specified Outcome: Number of Participants Experiencing Serious Adverse Events Within 30 Days
Description: Serious adverse events and adverse events related to the procedure and/or ablation catheter through 30 days post index ablation. This excludes the events identified in the primary safety endpoint.
Time Frame: 30 days
Population: Population includes all subjects with ablation catheter inserted.
Measure: Count of Participants; unit: Participants
Arm/Group | TactiCath SE
Number analyzed (Participants) | 151
Participants
  Serious AE Related to Device or Procedure | 5
  Non-Serious AE Related to Device or Procedure | 23

6. Other Pre Specified Outcome: Number of Participants Experiencing a Serious Adverse Event Within 1 Year
Description: Serious adverse events and adverse events related to the procedure and/or ablation catheter through 1 year post index ablation
Time Frame: 1 year
Population: Subjects with TactiCath SE inserted into vasculature
Measure: Count of Participants; unit: Participants
Groups:
- TactiCath SE: Catheter ablation with the TactiCath SE ablation catheter to achieve pulmonary vein isolation.
  TactiCath SE inserted
Arm/Group | TactiCath SE
Number analyzed (Participants) | 151
Participants
  Serious AE Related to Device or Procedure | 5
  Non-Serious AE Related to Device or Procedure | 23

7. Other Pre Specified Outcome: One-year Freedom From AF
Description: One-year freedom from AF, defined as freedom from symptomatic AF, atrial flutter (AFL), and atrial tachycardia (AT) lasting longer than 30 seconds through 9 months of follow-up after a 3-month blanking period.
Time Frame: 1 year
Population: Includes subjects with the following:
  * device inserted
  * RF energy delivered
  * Had 12M visit or failed endpoint
Measure: Count of Participants; unit: Participants
Arm/Group | TactiCath SE
Number analyzed (Participants) | 133
Participants | 108
Statistical Analysis 1: Comparison: TactiCath SE; Kaplan Meier Estimate of freedom from recurrence; Test type: Other; Kaplan-Meier Survival Estimate = 82.2, 95% CI 2-sided [74.7 to 87.6] — Kaplan-Meier estimate of freedom from recurrence at 1-year

8. Other Pre Specified Outcome: One-year Drug-free Success From AF
Description: One-year drug-free success defined as freedom from any AF/AFL/AT lasting at least 30 seconds or any Class I or III AAD after removal from antiarrhythmic drug therapy as assessed from the end of the 3-month blanking period to 12 months following the ablation procedure.
Time Frame: 1 year
Population: The analysis population included the following subjects:
  * Device inserted
  * Radiofrequency energy applied
  * 12M visit complete or failed endpoint
Measure: Count of Participants; unit: Participants
Groups:
- TactiCath SE Drug-Free Success Population: Catheter ablation with the TactiCath SE ablation catheter to achieve pulmonary vein isolation.
  TactiCath SE: Ablation to achieve pulmonary vein isolation.
  Includes all subjects with catheter inserted into vasculature.
Arm/Group | TactiCath SE Drug-Free Success Population
Number analyzed (Participants) | 136
Participants | 90
Statistical Analysis 1: Comparison: TactiCath SE Drug-Free Success Population; Kaplan-Meier estimate of freedom from recurrence or need for anti-arrhythmic medication; Test type: Other; Kaplan-Meier survival estimate = 68.2, 95% CI 2-sided [59.9 to 75.1]

9. Other Pre Specified Outcome: Changes in EQ-5D-5L Utility Scores
Description: Changes in EQ-5D-5L utility scores from baseline to follow up at 3, 6, and 12 months Utility scores range from 0 (worst) to 1 (best). A positive change indicates an improvement.
Time Frame: 1 year
Population: Subset of RF population with EQ-5D-5L data at both baseline and 12M
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RF Population
Number analyzed (Participants) | 71
score on a scale
  Change in EQ-5D-5L Utility from Baseline to 3M | 0.044 (0.108)
  Change in EQ-5D-5L Utility from Baseline to 6M: number analyzed (Participants) | 70
  Change in EQ-5D-5L Utility from Baseline to 6M | 0.066 (0.117)
  Change in EQ-5D-5L Utility from Baseline to 12M: number analyzed (Participants) | 65
  Change in EQ-5D-5L Utility from Baseline to 12M | 0.032 (0.158)

10. Other Pre Specified Outcome: Changes in AFEQT Scores
Description: Changes in AFEQT scores from baseline to follow up at 3, 6, and 12 months AFEQT scores range from 0 (most severe symptoms) to 100 (no limitation or disability). A positive change indicates an improvement in AF condition.
Time Frame: 1 year
Population: Subjects in RF population with available AFEQT data at both baseline and 12M
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RF Population
Number analyzed (Participants) | 71
score on a scale
  Change from Baseline to 3M | 25.8 (23.8)
  Change from Baseline to 6M: number analyzed (Participants) | 70
  Change from Baseline to 6M | 25.2 (21.9)
  Change from Baseline to 12M: number analyzed (Participants) | 66
  Change from Baseline to 12M | 29.1 (23.0)

11. Other Pre Specified Outcome: Health Care Utilization
Description: Cardiovascular-related health care utilization through 12 months post index ablation Cardiovascular-related health care utilization would include any office visits, tests, hospitalizations, or other interventions outside of routine follow up.
Time Frame: 1 year
Population: Subjects with device inserted and healthcare utilization data reported
Measure: Number; unit: Encounters
Arm/Group | TactiCath SE
Number analyzed (Participants) | 28
Encounters | 37

12. Other Pre Specified Outcome: Force Time Integral (FTI)
Description: Mean force-time integral across lesions for a subject FTI for a lesion is the product of contact force in grams and duration of radiofrequency ablation in seconds. The mean value for this product across all lesions for a subject is then calculated.
Time Frame: 0 days
Population: Subjects from RF population with FTI or LSI data available
Measure: Mean (Standard Deviation); unit: gram-seconds
Arm/Group | RF Population
Number analyzed (Participants) | 144
gram-seconds | 161.7 (103.7)

13. Other Pre Specified Outcome: Average Catheter Temperature
Description: This outcome is the average temperature (by lesion) for a case.
Time Frame: 0 days
Population: The population includes only subjects with at least some radiofrequency energy delivered.
Measure: Median (Inter-Quartile Range); unit: degrees celsius
Arm/Group | RF Population
Number analyzed (Participants) | 149
degrees celsius | 33.4 [32.5 to 34.6]

14. Other Pre Specified Outcome: Number of Participants With Recommended Irrigation Flow Rate Used During Procedure
Description: This outcome is whether or not the recommended irrigation flow rate was used for a case.
Time Frame: 0 days
Population: The population includes only subjects with at least some radiofrequency energy delivered.
Measure: Count of Participants; unit: Participants
Arm/Group | RF Population
Number analyzed (Participants) | 150
Participants | 140

15. Other Pre Specified Outcome: Contact Force During Procedure
Description: This outcome is the average contact force for a case.
Time Frame: 0 days
Population: The population includes only subjects with at least some radiofrequency energy delivered.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | RF Population
Number analyzed (Participants) | 149
grams | 12.1 (4.7)

16. Other Pre Specified Outcome: Total Procedure Time
Description: This outcome is the total procedure time for a case.
Time Frame: 0 days
Population: The population includes only subjects with at least some radiofrequency energy delivered.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | RF Population
Number analyzed (Participants) | 150
minutes | 159.5 [123.0 to 206.0]

17. Other Pre Specified Outcome: Ablation Time - First to Last Ablation
Description: This outcome is the total ablation time for a case. This is the time from first to last ablation.
Time Frame: 0 Days
Population: The population includes only subjects with at least some radiofrequency energy delivered.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | RF Population
Number analyzed (Participants) | 150
minutes | 84.0 [56.0 to 127.0]

18. Other Pre Specified Outcome: Fluoroscopy Time
Description: This outcome is the total fluoroscopy time for a case.
Time Frame: 0 days
Population: The population includes only subjects with at least some radiofrequency energy delivered.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | RF Population
Number analyzed (Participants) | 150
minutes | 9.0 [5.0 to 16.0]

19. Other Pre Specified Outcome: Radiofrequency (RF) Application Time
Description: This outcome is the total RF application time for a case.
Time Frame: 0 days
Population: The population includes only subjects with at least some radiofrequency energy delivered.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | RF Population
Number analyzed (Participants) | 149
minutes | 35.7 [28.9 to 51.9]

20. Other Pre Specified Outcome: Number of Participants Using AutoMark
Description: This outcome is the number of cases using AutoMark.
Time Frame: 0 days
Population: The population includes only subjects with at least some radiofrequency energy delivered.
Measure: Count of Participants; unit: Participants
Arm/Group | RF Population
Number analyzed (Participants) | 150
Participants | 149

21. Other Pre Specified Outcome: Lesion Index (LSI)
Description: Mean lesion index (LSI) across lesions by subject
  Lesion index is a proprietary score calculated as a function of power, contact force, and duration for a radiofrequency (RF) energy application. Scores start at 0 (no ablation) and do not have an upper limit. Applications must be at least 6 seconds in duration to generate a score. Lesion index is intended to provide feedback to the operator during an RF application.
Time Frame: 0 days
Population: Subjects from RF population with some LSI data available
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RF Population
Number analyzed (Participants) | 144
units on a scale | 4.3 (0.8)

ADVERSE EVENTS:
Time Frame: 30 days
Description: Adverse events include events that are not necessarily related to the device or procedure.
Arm/Group | TactiCath SE
All-Cause Mortality (participants affected / at risk) | 0/156
Serious Adverse Events (participants affected / at risk) | 21/156
Other Adverse Events (participants affected / at risk) | 25/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TactiCath SE (N=156)
Arrhythmias (Cardiac disorders) | 7 (8)
Atrial-Esophageal Fistula (Gastrointestinal disorders) | 1 (1)
Cardiac Perforation/Tamponade (Cardiac disorders) | 2 (2)
Cerebrovascular Accident/ Stroke (Nervous system disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Gastroparesis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Infections (Gastrointestinal disorders) | 1 (1)
Infections (Infections and infestations) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 3 (3)
Pericarditis (Cardiac disorders) | 1 (1)
Syncope/Dizziness (General disorders) | 1 (1)
Thromboembolism (Vascular disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Vascular Bleeding/Local Hematomas/Ecchymosis (Blood and lymphatic system disorders) | 1 (1)
Vascular Damage (Vascular disorders) | 1 (1)
Ventricular Tachyarrhythmia (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TactiCath SE (N=156)
Allergic Reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Chest Pain/Discomfort (Cardiac disorders) | 5 (5)
Epigastric Fullness (Gastrointestinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Infections (Infections and infestations) | 3 (3)
Infections (Renal and urinary disorders) | 1 (1)
Low Grade Temp (General disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 6 (6)
Syncope/Dizziness (Cardiac disorders) | 1 (1)
Vascular Access Complication (Vascular disorders) | 2 (2)
Vascular Bleeding/Local Hematomas/Ecchymosis (Vascular disorders) | 3 (3)
Volume Overload (Vascular disorders) | 2 (2)
Wrist Pain With Swelling And Bruising (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/63/NCT03354663/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/63/NCT03354663/SAP_001.pdf